CLINICAL TRIAL: NCT03099850
Title: Prospective Evaluation of Chronic Pancreatitis for Epidemiologic and Translational Studies - PROCEED Study
Brief Title: Prospective Evaluation of Chronic Pancreatitis for Epidemiologic and Translational Studies
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Institutes of Health (NIH) (NIH); University of Minnesota (Other); Ohio State University (Other); Baylor College of Medicine (Other); Indiana University (Other); University of Florida (Other); Cedars-Sinai Medical Center (Other); Stanford University (Other); Mayo Clinic (Other); University of Pittsburgh Medical Center (Other); Kaiser Permanente (Other)
Responsible Party: Sponsor
Other Study IDs: PA17-0104 (2020-1058); 1U01DK108328-01 (NIH); 2020-1058 (Other: MD Anderson Cancer Center); NCI-2021-00441 (Other: NCI-CTRP Clinical Trials Registry); NCT04753255 (obsolete NCT alias)
Record Dates: First submitted 2017-03-15; First posted 2017-04-04 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Pancreatitis
Keywords: Chronic Pancreatitis; Data management; Regulatory compliance; Protocol monitoring
MeSH Terms: conditions — Pancreatitis; Pancreatitis, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational cohort study of adult patients with suspected or definite CP: * Chronic Upper Abdominal Pain of Suspected Pancreatic Origin
  * Suspected Chronic Pancreatitis (Patients with Acute Pancreatitis, Recurrent Acute Pancreatitis, or Indeterminate CP without prior AP)
  * Definite Chronic Pancreatitis
  * Chronic Abdominal Pain- Undifferentiated Group
  Interventions: Other: Data Management and Monitoring

INTERVENTIONS:
Other: Data Management and Monitoring — The Coordinating and Data Management Center (CDMC) at MD Anderson Cancer Center responsible for monitoring protocol and regulatory compliance for consortium. CDMC responsible for maintaining and tracking IRB approval and regulatory documents from each site throughout the life of the study.
  * Study participants will complete questionnaires at baseline and during yearly follow-up. In the event a participant does not complete all or part of the patient or coordinator questionnaire, the study coordinator will complete questions via medical record review (e.g., demographics and family history) or via a telephone interview.
  * Biospecimen collection: blood, urine, saliva, stool. Biospecimens will be collected and processed in accordance with the CPDPC specimen collection procedures.
  * EUS or EGD with pancreatic fluid collection
  * imaging studies performed at baseline and at follow-up.
    * IV contrast-enhanced MRI and MRCP with secretin
    * IV contrast-enhanced CT Scan abdomen

SUMMARY:
The Coordinating and Data Management Center (CDMC) at MD Anderson Cancer will be responsible for the coordination and data management for the Prospective Evaluation of Chronic Pancreatitis for Epidemiologic and Translational Studies (PROCCEED) Study, which is part of the NIH U01 funded Consortium for the Study of Chronic Pancreatitis, Diabetes, and Pancreatic Cancer (CPDPC). No patient enrollment will occur at MDACC. All patient recruitment will occur at external sites that are a part of the CPDPC. The data management systems, auditing, and monitoring effort are supported by the MD Anderson Cancer Center Clinical Research Support Center (CRSC).

PROCEED is the first study in the USA that is carefully following participants to better understand factors that may be responsible for causing pancreatitis and how it progresses. The study is being conducted at the following 9 major clinical centers across the US:

* Baylor College of Medicine
* Cedars-Sinai Medical Center
* University of Florida
* Indiana University
* Mayo Clinic
* University of Minnesota
* Ohio State University
* Stanford University
* University of Pittsburgh

The study is enrolling participants who are at different stages of chronic pancreatitis, including those with no known pancreas disease (controls), and those with abdominal pain, one or more attacks of pancreatitis, or chronic pancreatitis. After enrollment, participants with abdominal pain and pancreatitis are asked to follow-up every year to learn about their symptoms and any changes in the disease. PROCEED investigators plan to use the detailed information they collect to better understand the disease and identify new treatments.

"More details and updated information about this study can be found at the study's public website: https://www.cpdpc-research-consortium.org/research- study-cpdpc-16-02-proceed".

ELIGIBILITY:
Inclusion Criteria:

1. Participants with chronic pancreatitis.

Exclusion Criteria:

ALL GROUPS EXCEPT GREEN GROUP I:

1. History of autoimmune or traumatic pancreatitis, or sentinel attack of acute necrotizing pancreatitis which results in suspected
2. Primary pancreatic tumors - pancreatic ductal adenocarcinoma, suspected cystic neoplasm (>1 cms in size or main duct involvement), neuroendocrine tumors, and other uncommon tumors.
3. Pancreatic metastasis from other malignancies.
4. History of solid organ transplant, HIV/AIDS.
5. Known isolated pancreatic exocrine insufficiency (e.g. in the absence of any eligible inclusion criteria).
6. Participants must not have medical or psychiatric illnesses or ongoing substance abuse that in the investigator's opinion would compromise their ability to tolerate study interventions or participate in longitudinal follow up.
7. Patients with known abnormal creatinine (GFR < 30) or renal failure (applies to patients with chronic upper abdominal pain of suspected pancreatic origin and suspected CP (Yellow) subgroups).
8. Failure to agree for longitudinal follow-up.
9. Known Pregnancy. All participants of childbearing potential, except if post-menopausal [i.e. no menses for ≥2 years] or had a hysterectomy, bilateral tubal ligation/clip (surgical sterilization) or surgical removal of both the ovaries), must have a negative urine or serum B-HCG pregnancy test documented within 2 days prior to any endoscopic or radiologic procedures done for research purposes. Any standard of care tests will follow institutional policies regarding pregnancy test.
10. Currently incarcerated.
11. Inability to get MRI/MRCP in patients with chronic abdominal pain of suspected pancreatic origin (Green II) or Suspected CP (Yellow groups) at baseline (e.g. metal object in the body which precludes performance of MRI).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants recruited from external sites.
Sampling Method: Non-Probability Sample
Enrollment: 2345 (Estimated)
Dates: Start 2017-02-28 (Actual); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs). Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | Through study completion; an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Li Liang, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Yadav D, Askew RL, Palermo T, Li L, Andersen DK, Chen M, Fisher WE, Fogel EL, Forsmark CE, Hart PA, Othman MO, Pandol SJ, Park WG, Topazian MD, Van Den Eeden SK, Vege SS, Yang Y, Serrano J, Conwell DL; Consortium for the Study of Chronic Pancreatitis, Diabetes; Pancreatic Cancer (CPDPC). Association of Chronic Pancreatitis Pain Features With Physical, Mental, and Social Health. Clin Gastroenterol Hepatol. 2023 Jul;21(7):1781-1791.e4. doi: 10.1016/j.cgh.2022.09.026. Epub 2022 Oct 1. PMID 36191836
- [Derived] Tirkes T, Yadav D, Conwell DL, Territo PR, Zhao X, Persohn SA, Dasyam AK, Shah ZK, Venkatesh SK, Takahashi N, Wachsman A, Li L, Li Y, Pandol SJ, Park WG, Vege SS, Hart PA, Topazian M, Andersen DK, Fogel EL; Consortium for the Study of Chronic Pancreatitis, Diabetes, Pancreatic Cancer (CPDPC). Quantitative MRI of chronic pancreatitis: results from a multi-institutional prospective study, magnetic resonance imaging as a non-invasive method for assessment of pancreatic fibrosis (MINIMAP). Abdom Radiol (NY). 2022 Nov;47(11):3792-3805. doi: 10.1007/s00261-022-03654-7. Epub 2022 Aug 29. PMID 36038644
- [Derived] Hart PA, Yadav D, Li L, Appana S, Fisher W, Fogel E, Forsmark CE, Park WG, Pandol S, Topazian MD, Van Den Eden SK, Vege SS, Bradley D, Serrano J, Conwell DL; Consortium for the Study of Chronic Pancreatitis, Diabetes, and Pancreatic Cancer (CPDPC). High Prevalence of Osteopathy in Chronic Pancreatitis: A Cross-sectional Analysis From the PROCEED Study. Clin Gastroenterol Hepatol. 2022 Sep;20(9):2005-2013. doi: 10.1016/j.cgh.2021.09.026. Epub 2021 Sep 24. PMID 34571258
- See also: MD Anderson Cancer Center — http://www.mdanderson.org